CLINICAL TRIAL: NCT01566591
Title: A Prospective, Double Blind, Randomized, Controlled Trial to Evaluate the Safety and Efficacy of the H1-Coil Deep Transcranial Magnetic Stimulation (TMS) in Conjunction With Mood Stabilizers in Subjects With Bipolar Depression
Brief Title: Safety and Efficacy Study of Deep Transcranial Magnetic Stimulation in Bipolar Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR-BIP-03
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2020-01

CONDITIONS: Bipolar Depression
Keywords: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Treatment (Sham Comparator): In the sham treatment,the electrical field induced by the sham coil cannot invoke any action potentials and if no action potentials are induced, then the electric field is insignificant and there is no treatment effect on the brain.
  Interventions: Device: Sham Treatment
- Deep TMS Treatment (Active Comparator): Deep TMS treatment is a new form of TMS which allows direct stimulation of deeper neuronal pathways than the standard TMS. The H-coil is a novel DTMS coil designed to allow deeper brain stimulation without a significant increase of electric fields induced in superficial cortical regions.
  Interventions: Device: Deep TMS Treatment

INTERVENTIONS:
Device: Deep TMS Treatment — 24 TMS treatments over 6 weeks .
  Arms: Deep TMS Treatment
Device: Sham Treatment — 24 TMS treatments over 6 weeks
  Arms: Sham Treatment

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of H1-Coil deep brain rTMS in subjects with bipolar depression, taking mood stabilizers and previously unsuccessfully treated with antidepressant medications.

DETAILED DESCRIPTION:
This is a multi center, randomized, double blind study to evaluate the efficacy and safety of H1-Coil deep brain rTMS in subjects with bipolar depression, taking mood stabilizers and previously unsuccessfully treated with antidepressant medications. The study is designed for a period of 8 weeks of which up to 3 weeks subjects will be tapered down from their medications and treated for 5 weeks. Two follow up visits will be performed at week 6 and 8 after the last TMS treatment. Mood and mental status will be closely monitored with standard psychological scales and assessments

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* patients suffering from an episode of bipolar depression (BP1 or BP2) according to DSM IV, with the additional requirement of duration for the current episode ≥ 4 weeks and CGI ≥ 4.
* Men and Women Ages 22-68 years.
* Negative answers on safety screening questionnaire for transcranial magnetic stimulation.
* Taking mood stabilizing medication (e.g., Lithium, Lamictal, Tegretol, Topamax, etc.) at a therapeutic dose or atypical antipsychotic medication which was prescribed as mood stabilizers by their treating physician, except for Leponex (Clozapine). According to the treating physician the patient is compliant with taking the mood-stabilizing medication.

Exclusion Criteria:

* patients suffering from other diagnoses on axis 1 such as schizophrenia , or suffering from psychotic depression in current episode.
* Diagnosed as suffering from Severe Borderline Personality Disorder or hospitalized due to exacerbation related to of borderline personality disorder. Subjects suffering from any other Severe Personality Disorder will also be excluded.
* Present suicidal risk as assessed by the investigator
* Patients with a bipolar cycle of less than 30 days.
* History of epilepsy or seizure (EXCEPT those therapeutically induced by ECT ) or history of such in first degree relatives.
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or history of significant head trauma with loss of consciousness for greater than or equal to 5 minutes.
* History of head injury.
* History of any metal in the head (outside the mouth).
* Metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or implanted medical pumps.
* Hearing loss.
* Individuals with a significant neurological disorder or insult including, but not limited to:

  * Any condition likely to be associated with increased intracranial pressure
  * Space occupying brain lesion
  * History of cerebrovascular accident
  * Transient ischemic attack within two years
  * Cerebral aneurysm
  * Dementia
  * Parkinson's disease
  * Huntington's chorea
  * Multiple sclerosis
* Current History of substance abuse including alcoholism or history of substance abuse including alcoholism within the past 6 months (except nicotine and caffeine).
* Inadequate communication with the patient.
* Under custodial care.
* Participation currently in another clinical study or enrolled in another clinical study within 30 days prior to this study.
* Participants who suffer from an unstable physical disease such as high blood pressure or acute, unstable cardiac disease
* Use of fluoxetine within 6 weeks of the baseline visit
* Use of a Monoamine Oxidase Inhibitor (MAOI) within 2 weeks of the baseline visit
* Current use of antidepressant medications during the course of the trial.
* Current use of Leponex (Clozapine).
* Previous treatment with TMS
* Women who are breast-feeding
* Known or suspected pregnancy
* Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.

Ages: 22 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-05; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
HDRS-21 Score measured by change from baseline. | 6 weeks from baseline

SECONDARY OUTCOMES:
Clinical antidepressant remission rate at the 6-week visit | 6 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yechiel Levkovitz, MD, Principal Investigator — Shalvata Mental Health Center
Locations (13):
- United States (9):
  - Advanced Mental Health Care Inc. - Juno Beach, Juno Beach, Florida
  - Advanced Mental Health Care Inc. - Palm Beach, Palm Beach, Florida
  - Advanced Mental Health Care Inc. - Royal Palm Beach, Royal Palm Beach, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Premier Psychiatric Group, Lincoln, Nebraska
  - Mount Sinai Hospital, New York, New York
  - Medical Uni. Of South Carolina (MUSC), Charleston, South Carolina
  - Senior Adults Specialty Research, Austin, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
- Center for Addiction and Mental Health (CAMH), Toronto, Ontario, Canada
- Klinik für Psychiatrie und Psychotherapie, Ludwig-Maximilians-Universität, Munich, Germany
- Israel (2):
  - Beer Yaacov Mental Health Center, Beer Yaacov
  - Lev Hasharon, Netanya